CLINICAL TRIAL: NCT04105881
Title: Correlation Between B Regulatory Cell and Vitamin D Status in Term and Preterm Labor
Brief Title: Correlation Between Vitamin D and B Regulatory Cell in Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Haitham Mohamed Sedky, Principle investigator, Assiut University
Other Study IDs: Dear
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Labor, Premature
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Contact Tracing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Total blood and serum

GROUPS / COHORTS (3):
- Full term labor: Measured by flow cytometry and ELUSA
  Interventions: Dietary Supplement: Investigation
- Preterm labor: Measured by flow cytometry and ELISA
  Interventions: Dietary Supplement: Investigation
- Control: For comparison
  Interventions: Dietary Supplement: Investigation

INTERVENTIONS:
Dietary Supplement: Investigation — Cross sectional intervention

SUMMARY:
During pregnancy , the maternal immune system is always confronted with fetal alloantigens. the immunological mechanisms that prevent the rejection of the fetus are still not under understood.

DETAILED DESCRIPTION:
During pregnancy , the maternal immune system is always confronted with fetal alloantigens. the immunological mechanisms that prevent the rejection of the fetus are still not under understood.the fetus is normally accepted by the maternal immune system despite despite the expression of paternal alloantigens. Normally, the fetus grows and develops very well with ongoing pregnancy.

B regulatory cells are increased in pregnant women compared to non-pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* healthy female according to the required groups

Exclusion Criteria:

* patient with infectious disease , tuberculosis ,tumor ,hematologic disease,metabolic bone disease or any other connective tissue diseases were excluded.
* Patient with viral hepatitis.
* serological evidence of HIV infection.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female Patient should be informed before sampling
Study Population: Healthy term delivery women and preterm labor women
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-02-10 (Estimated); Primary Completion 2020-03-10 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
Changes in number of B regulatory cell in pregnant woman | 9 months
  Immune system immunosuppressed to maintain fetus

CONTACTS AND LOCATIONS:
Overall Officials: khalid Hassanein, Principal Investigator — Microbiology and immunology department
Locations (2):
- Egypt (2):
  - Assiut university, Asyut, Asyut Governorate
  - Assiut university, Asyut

IPD SHARING:
Plan to Share IPD: Undecided
Role of immune system in maintenance of pregnancy

REFERENCES:
- [Result] Zahran AM, Zharan KM, Hetta HF. Significant correlation between regulatory T cells and vitamin D status in term and preterm labor. J Reprod Immunol. 2018 Sep;129:15-22. doi: 10.1016/j.jri.2018.07.004. Epub 2018 Jul 18. PMID 30029057
- [Result] Lima J, Martins C, Leandro MJ, Nunes G, Sousa MJ, Branco JC, Borrego LM. Characterization of B cells in healthy pregnant women from late pregnancy to post-partum: a prospective observational study. BMC Pregnancy Childbirth. 2016 Jun 6;16(1):139. doi: 10.1186/s12884-016-0927-7. PMID 27267973